CLINICAL TRIAL: NCT00311688
Title: An Omnibus Proleukin (IL-2) Trial in HIV Infected Patients Including Interrupted Versus Continuous Antiretrovirals (OPTICA)
Brief Title: Umbrella Study for HIV Infected Adults Enrolled in NIAID-Funded Interleukin-2 Studies
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRP 030/OPTICA; 10476 (Registry Identifier: DAIDS ES); IRP 030; OPTICA; NCT00359749 (obsolete NCT alias)
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: IL-2; Immunomodulatory Therapies
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (1):
- 1: Individuals will follow the schedule of the study they are participating in
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Biological response modifier in liquid form; dosage of drug will vary by study
  Other Names: IL-2

SUMMARY:
Interleukin-2 (IL-2) is a protein found naturally in the blood that helps boost the immune system. The purpose of this study is to provide long-term treatment and monitoring of HIV infected people enrolled in NIAID-funded studies investigating the use of laboratory-made IL-2 for the treatment of HIV infection.

DETAILED DESCRIPTION:
IL-2 is a biological response modifier that can improve the body's response to disease. It is hoped that IL-2 treatment can help restore CD4 cell counts and immune function in people whose immune systems have been damaged by HIV. Over the last 10 years, NIAID has sponsored a number of important studies of IL-2 in HIV infected people; many of these trials are ongoing. This study was developed in an effort consolidate these separate, smaller trials into one larger study so that results between the trials can be shared and used to develop future protocols. This study is an umbrella study that will provide long-term administrative support, treatment, and monitoring for ongoing Phase I and II IL-2 trials and their participants. It is primarily intended for patients in the extension phases of any previous NIAID Clinical Center HIV Program (NIAID/CCMD) intramural research protocols in which IL-2 therapy continues to be offered. Blood collection will occur through a patient's participation in this study.

Participants will continue to follow the protocol in which they originally enrolled. A desired therapeutic goal or "CD4 plateau" will be used in most cases to help clinicians determine when a participant requires additional IL-2. In general, if a participant has two or more consecutive CD4 counts below the CD4 plateau, additional IL-2 will be administered to that patient. In maintaining uniformity among the many trials being consolidated under this trial, the frequency and nature of study visits will be solely dictated by this umbrella study. Participants will also be asked to join an optional substudy: Interrupted Versus Continuous Antiretrovirals Involving Randomization from the Umbrella Study (ICARUS).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Current participation and presently in good standing in a NIAID/CCMD clinical trial involving the use of IL-2 for the treatment of HIV-1 infection. Additional HIV-1 infected people who are IL-2 naive may be selected by the investigator for this study.
* Willing to take antiretrovirals within a 10-day period surrounding each IL-2 cycle. Individual protocols may be modified as needed by the investigator to permit IL-2 therapy in the absence of antiretrovirals.
* Willing to accept additional IL-2 therapy when needed
* Willing to use acceptable forms of contraception during a minimum 10-day period surrounding each IL-2 injection

Exclusion Criteria:

* History of noncompliance with prior NIAID/CCMD protocols
* Any organic central nervous system (CNS) abnormality requiring treatment with antiseizure medication
* Unless previously exempted for this requirement, current or history of Crohn's disease, psoriasis, or other autoimmune or inflammatory disease with potentially life-threatening complications
* Significant heart, lung, kidney, rheumatologic, gastrointestinal, or CNS disease that may pose an unacceptable risk to the participant during IL-2 therapy
* Psychiatric illness that, in the opinion of the investigator, may interfere with the study
* Current or recent substance abuse that, in the opinion of the investigator, may interfere with the study
* Refuse to follow Clinical Center policy on partner notification
* History of optic neuritis
* Refuse to allow extra blood specimens to be stored for potential use in future studies of HIV-1 infection or the immune system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
CD4 counts in participants treated with IL-2 and discontinued antiretroviral therapy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Davey, Jr., MD, FACP, Study Chair — NIAID HIV Research Clinic, Laboratory of Immunoregulation, NIAID
Locations (1):
- NIH Intramural Research Program ACTG CRS, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anaya JP, Sias JJ. The use of interleukin-2 in human immunodeficiency virus infection. Pharmacotherapy. 2005 Jan;25(1):86-95. doi: 10.1592/phco.25.1.86.55629. PMID 15767224
- [Background] Marchetti G, Franzetti F, Gori A. Partial immune reconstitution following highly active antiretroviral therapy: can adjuvant interleukin-2 fill the gap? J Antimicrob Chemother. 2005 Apr;55(4):401-9. doi: 10.1093/jac/dkh557. Epub 2005 Feb 24. PMID 15731201
- [Background] Temesgen Z. Interleukin-2 for the treatment of human immunodeficiency virus infection. Drugs Today (Barc). 2006 Dec;42(12):791-801. doi: 10.1358/dot.2006.42.12.1025703. PMID 17285152